CLINICAL TRIAL: NCT02537054
Title: Intravitreal Aflibercept (Eylea) for Therapy of Choroidal Neovascularization (CNV) and Fibrovascular Proliferation (FVP) in Patients With Pseudoxanthoma Elasticum (PXE)
Brief Title: Intravitreal Aflibercept for Therapy of Patients With Pseudoxanthoma Elasticum (PXE)
Acronym: EyNeP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Frank G. Holz, Prof. Dr. med. Frank G. Holz, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUG-201202-EyNeP
Record Dates: First submitted 2015-08-21; First posted 2015-09-01 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: Choroidal neovascularization; Angioid streaks; Pseudoxanthoma Elasticum; vascular endothelial growth factor; aflibercept
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Choroidal Neovascularization; Angioid Streaks | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental): 2 mg/ dose (pro re nata, maximum 1 dose/ month), intravitreal use
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea

SUMMARY:
The purpose of this study is to determine whether Aflibercept (Eylea) is effective in the treatment of choroidal neovascularization and fibrovascular proliferation in patients with pseudoxanthoma elasticum (PXE) in terms of preservation or improvement of visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PXE by moleculargenetic diagnosis and/or skin biopsy
* Diagnosed CNV or FVP
* Age 18-65 years
* Voluntary participation in this study as proven by written informed consent
* Ability to follow study instructions and likely to attend and complete all required visits
* Best corrected visual acuity between 20/400 and 20/20 at treated eye
* Male and female patients with childbearing potential must use an approved contraceptive method (Pearl Index < 1) before and during the trial
* Pre-menopausal female patients with childbearing potential: a negative pregnancy test must be obtained

Exclusion Criteria:

* Subject is unable to understand the nature, scope, significance and consequences of this clinical trial
* Patients with known allergy or hypersensitivity to Eylea or preparations with similar chemical structure
* Treatment in another clinical trial with therapeutic intervention or use of any other investigational medicinal product (IMP) during the trial of within 30 days before enrolment
* Known or persistent abuse of medication, drugs or alcohol
* Women who are pregnant or breast feeding
* Lack of eligibility at discretion of the investigator
* Ocular operations within a month prior to enrolment
* Non-controlled glaucoma
* Active intraocular inflammation or inflammation of ocular adnexa
* Other diseases resulting in distinct visual constraint
* Distinct opacification of optical media
* Distinct subretinal fibrosis and /or atrophy that prevents a relevant treatment effect by Aflibercept at discretion of investigator
* Serious cardiovascular problems or stroke within 6 months before enrolment
* Simultaneous use of other Vascular Endothelial Growth Factor (VEGF)-inhibiting medication (systemic or ocular) within a month prior to enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Change in distance best corrected visual acuity between end-of study visit and screening visit | Screening visit (day -28 - 0) and end-of-study visit (day 360 +/- 7)

SECONDARY OUTCOMES:
Change in light increment sensitivity of central visual field between end-of study visit and screening visit measured by microperimetry | Screening visit (day -28 - 0) and end-of-study visit (day 360 +/- 7)
Change in chorioretinal neovascularization and leakage measured by angiography between end-of study visit and screening visit | Screening visit (day -28 - 0) and end-of-study visit (day 360 +/- 7)
Change in sub- and intraretinal und subpigmentepithelial fluids assessed using optical coherence tomography (OCT) | Screening visit (day -28 - 0) and end-of-study visit (day 360 +/- 7)
Extent of fibrovascular proliferation on optical coherence tomography (OCT) imaging | Screening visit (day -28 - 0) and end-of-study visit (day 360 +/- 7)
Changes fundus autofluorescence images using a confocal scanning laser ophthalmoscope (cSLO) | Screening visit (day -28 - 0) and end-of-study visit (day 360 +/- 7)
Occurence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 12 months
Change in the health status of the total population measured by quality of life questionnaire Visual Function Questionnaire (VFQ)-25 | Screening visit (day -28 - 0) and end-of-study visit (day 360 +/- 7)

CONTACTS AND LOCATIONS:
Overall Officials: Frank G. Holz, MD, DPhil, Principal Investigator — University Clinic Bonn
Locations (1):
- Department of Ophthalmology, Universtiy of Bonn, Bonn, Germany